CLINICAL TRIAL: NCT02508454
Title: The Miami Heart Study at Baptist Health South Florida: A Prospective Study of Sub-Clinical Cardiovascular Disease and Emerging Cardiovascular Risk Factors in Asymptomatic Young & Middle-Aged Adults
Brief Title: The Miami Heart Study at Baptist Health South Florida
Acronym: MiHEART
Status: Active, not recruiting | Type: Observational
Sponsor: Baptist Health South Florida (Other)
Collaborators: Quest Diagnostics-Nichols Insitute (Industry); University of California, Los Angeles (Other)
Responsible Party: Sponsor
Other Study IDs: 14-042
Record Dates: First submitted 2015-06-09; First posted 2015-07-27 (Estimated); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Cardiovascular Disease
Keywords: Prevention; Screening; Biobanking
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Approximately 115 mls of blood will be drawn by a Registered Nurse. Blood samples will be tested for markers of the diseases and health conditions under investigation. These will include standard markers (cholesterol, blood sugar, etc) and novel markers which are not commonly evaluated by a physician. Additionally, any remaining blood samples will be stored and kept for future risk factor evaluation, biomarker testing and genetic studies.
  Whole blood and serum will be retained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Greater Miami Area Community: Members of the Miami area who qualify for the study, are not an employee of BHSF, and enroll.
- Baptist Health South Florida Employees: Employees of BHSF who qualify for the study and enroll.

SUMMARY:
The Miami Heart Study at Baptist Health will be an observational, longitudinal and prospective cohort study in a target population of 4000 healthy subjects (40-65 years old) consisting of members from the Greater Miami Area (including eligible BHSF(Baptist Health South Florida) employees). Baseline examination will consist of (1) assessment for cardiovascular risk factors (including lifestyle and psychosocial factors); (2) screening for subclinical atherosclerosis using Coronary CT angiogram, Coronary Artery Calcium (CAC) testing, vascular 2D/3D ultrasound, endothelial function, arterial stiffness and (3) blood sampling for determination of traditional risk factors, advanced "omics" and biobanking. Participants will be followed yearly via telephone, email, or mail for change in health status with a focus on cardiovascular disease events, including acute myocardial infarction and other forms of coronary heart disease (CHD), stroke, and congestive heart failure; mortality; and for cardiovascular disease interventions.

The Miami Heart Study at Baptist Health is expected to identify new imaging and biological factors associated with the presence and feature of earliest markers of subclinical atherosclerotic disease and provide opportunities for discovery/validation of novel biomarkers to identify these high-risk features. This is expected to lead to advances in understanding of evolution and progression of atherosclerotic cardiovascular disease starts with an ultimate goal of establishing more personalized, evidence-based approach to medical care.

DETAILED DESCRIPTION:
What is this study about? The Miami Heart Study is a long term observational research study which is designed to identify new and novel relationships between risk factors, genetics, lifestyle behaviors and cardiovascular disease in the greater Miami area. Miami is uniquely situated to capture a diverse, multi-ethnic population. As an employee of Baptist Health and a very important stakeholder in Baptist Health's mission, you are being asked to take part in this research study. The investigators expect approximately 4,000 members of the South Florida community and/or employees of Baptist Health to participate in this study over the next 5 years.

The research study aims to better understand heart disease and what causes it. Heart disease often starts many years before a person has a heart attack or develops symptoms of heart disease. This is called subclinical disease - and it refers to heart disease and the body processes causing heart disease, at a stage before any symptoms are experienced. Although doctors and researchers have a good understanding of heart disease in some areas, subclinical disease is not very well understood.

Better understanding subclinical disease can allow doctors and healthcare staff to intervene and prevent the process from developing further and causing symptomatic (with symptoms) heart disease. Progression refers to the process by which subclinical (without symptoms) heart disease develops into clinical (with symptoms) disease.

Therefore, the purpose of this research study is to:

* To examine the presence and severity of subclinical disease in the South Florida community.
* To examine what unique factors contribute to development of subclinical disease and appearance of clinical symptoms.

In the future, the investigators hope this information will allow us to better predict and prevent the development heart disease in diverse populations. Participants will be asked to come to the Miami Heart Study clinic for an examination that may take 4 to 6 hours to complete. During the examination, information about the participant's health will be collected and standard procedures routinely done a physician's office such as height, weight, and blood pressure will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Current full time/part-time employees of BHSF (occupational cohort) or resident of Greater Miami Area for at least six months (community cohort)
* Age 40 to 65 years
* Asymptomatic individuals free of any known cardiovascular event
* Able to comprehend and sign an informed consent form

Exclusion Criteria:

* Prior history of major cardiovascular events (angina, myocardial infarction, prior coronary revascularization)
* History of cerebrovascular disease including stroke and transient ischemic attack (TIA)
* History of peripheral arterial disease (PAD)
* History of either diagnosis or surgery for Abdominal Aortic Aneurysm (AAA)
* Heart failure
* Weight greater than 350 lbs
* Any contraindication to CT scans or iodinated contrast
* Active treatment for cancer
* Currently pregnant, breastfeeding, or suspect they may be pregnant.
* Patients who do not agree to an informed consent

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Since the MiHEART Study is primarily concerned with the determinants and natural history of subclinical cardiovascular disease, participants with known clinical disease will not be recruited. Most exclusion criteria relate to the long-term nature of the study or to incompatibility with certain study procedures. Eligibility (or ineligibility) status will be determined from self-reported information.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2015-05 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in presence of subclinical cardiovascular disease burden among cohort as measured through yearly followup questionnaire. | Participants will be followed yearly for 5 years following completion of thier baseline visit.
  To assess and characterize the presence of subclinical cardiovascular disease burden among middle-aged asymptomatic individuals.
Change from baseline in severity of subclinical cardiovascular disease burden among cohort as measured through yearly followup questionnaire. | Participants will be followed yearly for 5 years following completion of thier baseline visit.
  To assess and characterize the severity of subclinical cardiovascular disease burden among middle-aged asymptomatic individuals.

SECONDARY OUTCOMES:
Associated cost savings of early discovery of disease. | Participants will be followed yearly for 5 years following completion of thier baseline visit.
  To develop population-based methods for characterizing cardiovascular risk among middle-aged asymptomatic persons as well cost effectiveness for such paradigms in appropriately resource allocation for early cardiovascular disease management.

CONTACTS AND LOCATIONS:
Overall Officials: Khurram Nasir, MD, MPH, Principal Investigator — Baptist Health South Florida
Locations (1):
- Raul Herrera, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ichikawa K, Ronen S, Bishay R, Krishnan S, Benzing T, Kianoush S, Aldana-Bitar J, Cainzos-Achirica M, Feldman T, Fialkow J, Budoff MJ, Nasir K. Coronary Plaque Volume in an Asymptomatic Population: Miami Heart Study at Baptist Health South Florida. JACC Cardiovasc Imaging. 2026 Jan;19(1):49-60. doi: 10.1016/j.jcmg.2025.08.001. Epub 2025 Sep 8. PMID 40920149
- See also: Miami Heart Study Website - English — http://miamiheartstudy.com/en/Pages/default.aspx
- See also: Miami Heart Study Website -Español — http://miamiheartstudy.com/sp/Paginas/inicio.aspx